CLINICAL TRIAL: NCT00173511
Title: Cardiovascular Events in Patients With CAD During Emergent Endoscopy for Upper Gastrointestinal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700701
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: 24 hr Holter monitor

SUMMARY:
Background:

Upper gastrointestinal (GI) bleeding, a common disorder encountered at emergency room, may cause hypotension and tachycardia that may in turn result in myocardial ischemia in patients with coronary artery disease (CAD). An emergent endoscopy with hemostasis is the mainstay of management. However, endoscopy itself may result in myocardial ischemia. Whether myocardial ischemia and arrhythmia occurs more frequently during emergent endoscopy in patients with CAD remains unknown.

Objective:

To determine whether the risk of myocardial ischemia and arrhythmia is increased during emergent endoscopy in patients with CAD.

Method:

Adult patients with documented CAD undergoing emergent endoscopy due to UGI bleeding are included. Adult patients without CAD undergoing emergent endoscopy due to UGI bleeding were included as the control group. The expected case numbers were 50 patients in each group. Patients with terminal illness, pregnancy, active lung disease requiring ventilator support are excluded. Before endoscopy, symptoms of myocardial ischemia, blood pressure, heart rate, O2 saturation, hemogram, baseline 12-lead EKG, and cardiac enzyme are obtained. All patients are monitored with Holter EKG since 10 minutes before endoscopy to 2 hours after the procedure. Blood pressure, heart rate, and O2 saturation are closely monitored during the procedure. Endoscopy is performed by experienced endoscopist and endoscopic hemostasis is done according to the types of lesions. The duration of endoscopy, types of endoscopic hemostasis, and blood pressure are recorded. After endoscopy, symptoms of myocardial ischemia, blood pressure, heart rate, O2 saturation, hemogram, baseline 12-lead EKG, and cardiac enzyme are checked again.

Keywords: Emergent endoscopy, coronary artery disease, cardiovascular events

DETAILED DESCRIPTION:
Expected Result and Implication If myocardial ischemia is not increased in CAD patients undergoing emergent endoscopy, then this technique can be used safely in this group of patients. If myocardial ischemia occurs more frequently in CAD patients undergoing emergent endoscopy, we can try to analyze factors associated with increased risk, such as duration of endoscopy, severity of anemia, or drugs used for endoscopic hemostasis. Then we can try to avoid these predisposing factors and increase the safety of emergent endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with documented CAD undergoing emergent endoscopy due to UGI bleeding are included.
* Adult patients without CAD undergoing emergent endoscopy due to UGI bleeding were included as the control group.

Exclusion Criteria:

* Acute coronary syndrome before enrollment
* Unable to receive upper endoscopy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Po Wang, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tseng PH, Liou JM, Lee YC, Lin LY, Yan-Zhen Liu A, Chang DC, Chiu HM, Wu MS, Lin JT, Wang HP. Emergency endoscopy for upper gastrointestinal bleeding in patients with coronary artery disease. Am J Emerg Med. 2009 Sep;27(7):802-9. doi: 10.1016/j.ajem.2008.06.018. PMID 19683108